CLINICAL TRIAL: NCT02485327
Title: An Open-label, 2 Replicate Single Dose Euglycemic Glucose-Clamp Trial to Characterize PK and PD Within-Subject Variability of a Single Dose of Afrezza Inhaled Technosphere Insulin in Patients With Diabetes Mellitus Type 1 (T1DM)
Brief Title: PK and PD Within-Subject Variability of a Single Dose of Afrezza Inhaled Technosphere Insulin in Patients With Diabetes Mellitus Type 1 (T1DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDY14329; 2015-001008-74 (EudraCT Number); U1111-1168-4442 (Other: UTN)
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Afrezza® (Experimental): Two-period, replicate single dose, euglycemic clamp study. There will be 2 treatment periods with a replicate administration of 1 dose of Afrezza TI (40U) in both periods.
  Each patient will be given a replicate administration of 1 dose level of Afrezza TI with washout duration between treatment periods (5-19 days between periods, ie, 7 to 21 days between dosing occasions).
  Interventions: Drug: Technosphere Insulin SAR439065 Afrezza®

INTERVENTIONS:
Drug: Technosphere Insulin SAR439065 Afrezza® — Pharmaceutical form: dry powder
  Route of administration: oral inhalation
  Other Names: Afrezza®

SUMMARY:
Primary Objective:

To characterize the within-subject variability in systemic exposure pharmacokinetic (PK) to insulin of a replicate single dose of Afrezza inhaled Technosphere Insulin (TI) in T1DM patients in a euglycemic clamp setting.

To characterize the within-subject variability in the metabolic activity (pharmacodynamic [PD]) of a replicate single dose of Afrezza inhaled TI in T1DM patients in a euglycemic clamp setting.

Secondary Objectives:

To assess the PK characteristics of a replicate single dose of Afrezza inhaled TI in a euglycemic clamp setting.

To assess the PD characteristics of a replicate single dose of Afrezza inhaled TI in a euglycemic clamp setting.

To assess the safety and tolerability of a replicate single dose of Afrezza inhaled TI in a euglycemic clamp setting.

DETAILED DESCRIPTION:
The maximum study duration per patient is approximately 9 weeks (screening of 3 to 28 Days, treatment period of 2 days [Periods 1 and 2], washout period of 5 to 19 days [between treatment period], and end-of-study visit of 7 to 14 days after study drug administration in Period 2).

ELIGIBILITY:
Inclusion criteria :

* Body weight between 50 and 95 kg, inclusive, body mass index between 18.5 and 29 kg/m², inclusive.
* Fasting serum C-peptide <0.3 nmol/L.
* Glycohemoglobin (HbA1c) ≤75 mmol/mol (≤9%).
* Stable insulin regimen for at least 2 months prior to study (with respect to safety of the patient and scientific integrity of the study).
* Certified as otherwise healthy for T1DM patient by assessment of medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculoskeletal system), unless the Investigator considers any abnormality to be clinically irrelevant and not interfering with the conduct of the study (with respect to safety of the subject and scientific integrity of the study).
* Normal vital signs after at least 10 minutes resting in supine position:

  * 95 mmHg <systolic blood pressure (SBP) <150 mmHg.
  * 45 mmHg <diastolic blood pressure (DBP) <95 mmHg.
  * 50 bpm <heart rate (HR) <90 bpm.
* Normal standard 12-lead electrocardiogram (ECG) after at least 10 minutes resting in supine position; 120 ms <PR <220 ms, QRS <120 ms, QTc ≤450 ms if male, ≤470 ms if female.
* Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for diabetes patients; however serum creatinine should be strictly below the upper laboratory norm; alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the patient has documented Gilbert syndrome) should not be above 1.5 x upper limit of normal (ULN).
* Women of childbearing potential (less than 2 years postmenopausal or not surgically sterile for more than 3 months), must have a negative serum beta-human chorionic gonadotropin (β-HCG) pregnancy test at screening and a negative urine β-HCG pregnancy test at Day 1 in all treatment periods (TPs) and must use a highly effective method of birth control, which is defined as those which result in a low failure rate (ie, less than 1% per year) according to the Note for guidance on nonclinical safety studies for the conduct of human clinical trials for pharmaceuticals (CPMP/ICH/286/95, modifications). During the entire study female subjects of childbearing potential must use 2 independent methods of contraception, eg, diaphragm and spermicide-coated condom. The use of a condom and spermicidal creams is not sufficiently reliable. For postmenopausal women with presence of less than 2 years post menopausal, and not surgically sterile for more than 3 months, the hormonal status will be determined (follicle-stimulating hormone [FSH] >30 IU/L).
* Having given written informed consent prior to undertaking any study-related procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national (German) laws in force relating to biomedical research.
* Not under any administrative or legal supervision.
* Nonsmoking at least for the last 6 months before screening (to be confirmed by serum cotinine <25 µg/L or urine <500 µg/L).
* Pulmonary function test at screening: forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) greater than or equal to 70% of the individual prediction according to the equation of the Third National Health and Nutrition Examination Survey (NHANES III).

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from T1DM), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Severe hypoglycemia resulting in coma/seizures or requiring assistance of another person, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 3 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day).
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* If female, pregnancy (defined as positive β-HCG blood test), breastfeeding at screening and before any treatment periods (defined as positive β-HCG urine test).
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or PD half-life of the medication, with the exception of insulin, stable treatment (at least 2 months) with thyroid hormones, lipid-lowering and antihypertensive drugs and if female with the exception of hormonal contraception or menopausal hormone replacement therapy.
* Any vaccination within the last 28 days.
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any patient in the exclusion period of a previous study according to applicable regulations.
* Any patient who cannot be contacted in case of emergency.
* Any patient who is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), antihepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, and cotinine).
* Positive alcohol test.
* Presence or history of any acute or chronic obstructive bronchopulmonary disease (COPD) including asthma, cancer.
* Upper respiratory tract infection within 8 weeks before screening.
* Known hypersensitivity to Afrezza TI and excipients.
* Inability, in the opinion of the Principal Investigator or a designee, to adequately inhale Afrezza powder.
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first-degree relatives (parents, siblings, or children).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameter: area under the serum insulin concentration time curve from time 0 to 8H (INS-AUC0-8H) | 8 hours
Assessment of PD parameter: area under the glucose infusion rate curve (GIR) necessary to maintain euglycemia during the euglycemic clamp over 8 hours | 8 hours

SECONDARY OUTCOMES:
Assessment of PK parameter: maximum Afrezza insulin serum concentration (INS-Cmax) | 8 hours
Assessment of PK parameter: time to INS-Cmax (INS-tmax) | 8 hours
Assessment of PD parameter: maximum smoothed GIR (GIRmax) | 8 hours
Assessment of PD parameter: time to GIRmax (GIR-Tmax) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Mainz, Germany